CLINICAL TRIAL: NCT04706585
Title: Thalassemia in Indonesia: Current Knowledge, Attitude, and Practice Among Young People
Brief Title: Thalassemia Knowledge in Young People of Indonesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Sponsor
Other Study IDs: MHS001
Record Dates: First submitted 2020-12-08; First posted 2021-01-13 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Thalassemia
Keywords: Thalassemia; Indonesia; Youth
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth: Young people in Indonesia between the age of 15-24 who are currently attending high school or university-level education to fill in our online survey.

SUMMARY:
There is still an ongoing lack of awareness about thalassemia among Indonesians despite high disease prevalence, and this is associated with poor implementation of preventive and promotive measures. Thalassemia experts argue that education and raising awareness about thalassemia must be done from an early age in order to relieve the heavy disease burden of thalassemia, especially in Indonesia as it is geographically located in the thalassemia belt. In spite of this, there has been limited research on public perception towards thalassemia in Indonesia, particularly among young people.

In this study, the researcher will ask young people in Indonesia between the age of 15-24 who are currently attending high school or university-level education to fill in an online survey. The survey consists of questions about the participants' demographic information as well as their knowledge, attitude, and practice (KAP) scores towards thalassemia. The study is expected to run from December 2020 to March 2021, with the online survey distributed in January 2021. Data collection will immediately follow, and it will be analyzed using univariate, bivariate, and multivariate analysis using the appropriate statistical tests. The findings gathered from this study will be vital in providing new insight into how the youth sees thalassemia in Indonesia. Such public health information will prove to be important in designing successful thalassemia intervention and education programs for Indonesian youth.

DETAILED DESCRIPTION:
Research concept

In this study, the researcher will ask young people in Indonesia between the age of 15-24 who are currently attending high school or university-level education to fill in an online survey. The survey consists of questions about the participants' demographic information as well as their knowledge, attitude, and practice (KAP) scores towards thalassemia. The study is expected to run from December 2020 to March 2021, with the online survey distributed in January 2021. Data collection will immediately follow, and it will be analysed using univariate, bivariate, and multivariate analysis using the appropriate statistical tests.

Study design

To evaluate the knowledge, attitude, and practice of Indonesian youth, the study design used will be observational, cross-sectional. An online questionnaire developed by the research team along with several experts is expected to be disseminated to the target population in January 2021. In light of the ongoing pandemic, this is expected to be a nationwide study where most of the work is done via online methods.

Place and period of study

This study will be conducted via online survey due to the ongoing pandemic situation. The study is expected to run from December 2020 to March 2021.

ELIGIBILITY:
Inclusion Criteria:

* Survey participants are based in Indonesia
* Survey participants are between the age of 15-24 and currently attending high school or university level education
* Survey participants include both thalassemia-affected patients and non-patients
* Survey participants have understood and given their consent for the research

Exclusion Criteria:

* Currently not studying/living in Indonesia
* Below the age of 15 or above 24
* No consent is given

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In this study, we will ask young people in Indonesia between the age of 15-24 who are currently attending high school or university-level education to fill in our online survey.
Sampling Method: Non-Probability Sample
Enrollment: 1010 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Indonesian youth's level of knowledge on thalassemia | Baseline, pre-intervention
  To determine the relationships among Indonesian youth's demographic, education and socioeconomic level to their knowledge of thalassemia via a validated self-developed questionnaire. Knowledge will be assessed through question of common knowledges surrounding thalassemia, a final score (out of 100) will be used as representation of knowledge level (0-25: poor, 25-50 moderate, 51-75 good, and 76-100 very good) will be evaluated after participants answer all the questions.
Indonesian youth's attitude towards thalassemia | Baseline, pre-intervention
  To determine the relationships among Indonesian youth's demographic, education and socioeconomic level to their attitude towards thalassemia via a validated self-developed questionnaire. (using a Likert scale of 1 to 4 - with 1 being "strongly agree" and 4 "strongly disagree")
Indonesian youth's practice towards thalassemia | Baseline, pre-intervention
  To determine the relationships among Indonesian youth's demographic, education and socioeconomic level to their action and practice towards prevention of thalassemia via a validated self-developed questionnaire. (using a Likert scale of 1 to 4 - with 1 being "strongly agree" and 4 "strongly disagree")

SECONDARY OUTCOMES:
Willingness to undergo thalassemia screening | Baseline, pre-intervention
  To determine Indonesian youth's willingness (using a Likert scale of 1 to 4 - with 1 being "strongly agree" and 4 "strongly disagree") to undergo thalassemia screening independently

CONTACTS AND LOCATIONS:
Overall Officials: Pustika A Wahidiyat, Professor., Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Mikhael Yosia, Dr., Principal Investigator — Fakultas Kedokteran Universitas Indonesia; Edward C Yo, Study Director — Fakultas Kedokteran Universitas Indonesia; Muhammad M Wildani, Study Chair — Fakultas Kedokteran Universitas Indonesia; Visabella R Triatmono, Study Chair — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Fakultas Kedokteran Universitas Indonesia - Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
We are not planning on making the IPD available for other researchers due to the current format of our informed consent.

REFERENCES:
- [Background] Marengo-Rowe AJ. The thalassemias and related disorders. Proc (Bayl Univ Med Cent). 2007 Jan;20(1):27-31. doi: 10.1080/08998280.2007.11928230. PMID 17256039
- [Background] Husna N, Sanka I, Arif AA, Putri C, Leonard E, Handayani NSN. Prevalence and distribution of thalassemia trait screening. J Med Sci. 2017 Jul;49(3):106-13.
- [Background] Wahidiyat PA, Sari TT, Rahmartani LD, Setianingsih I, Iskandar SD, Pratanata AM, et al. An insight into Indonesian current thalassaemia care and challenges. ISBT Sci Ser. 2020;15(3):334-41.
- [Background] Wahidiyat I, Wahidiyat PA. Genetic problems at present and their challenges in the future: thalassemia as a model. Paediatr Indones. 2006;46(5):189-94.